CLINICAL TRIAL: NCT03580148
Title: A Randomized Trial of Cortisone Injection Versus Bone Marrow Aspirate Injection Therapy for Glenohumeral Osteoarthritis
Brief Title: BMA vs Cortisone for Glenohumeral Osteoarthritis
Acronym: BMAC
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Women's College Hospital (Other)
Collaborators: University of Toronto (Other)
Responsible Party: Principal Investigator, Dr. Tim Dwyer, Dr. Tim Dwyer, Orthopaedic Surgeon, Principal Investigator, Women's College Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015-0069-B
Record Dates: First submitted 2018-06-22; First posted 2018-07-09 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Osteo Arthritis Shoulders
Keywords: osteoarthritis; glenohumeral joint; arthritis; shoulder
MeSH Terms: conditions — Osteoarthritis; Arthritis | interventions — Cortisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cortisone (Active Comparator): Patients randomized to this arm will receive one (1) ultrasound guided injection of 80mg Depo Medrol cortisone in the glenohumeral joint of the affected shoulder. Procedure time of approximately 10 minutes
  Interventions: Drug: Cortisone
- Bone Marrow Aspirate (Active Comparator): Patients randomized to this arm will receive one (1) ultrasound injection of bone marrow aspirate, harvested from the posterior superior iliac spine, and injected into the glenohumeral joint of the affected shoulder. Procedure time of approximately 45 minutes
  Interventions: Biological: Bone Marrow Aspirate

INTERVENTIONS:
Drug: Cortisone — Patients randomized to receive this study intervention will undergo one ultrasound guided 80mg Depo Medrol GHJ injection
  Other Names: 00030767 DEPO-MEDROL 80 MG/ML
  Arms: Cortisone
Biological: Bone Marrow Aspirate — Patients randomized to receive this study intervention will have, under sterile conditions and after injection of local anesthetic, 10 mls of bone marrow aspirate taken from the posterior superior iliac spine and injected under ultrasound guidance to the glenohumeral joint
  Other Names: BMA
  Arms: Bone Marrow Aspirate

SUMMARY:
This randomized trial seeks to investigate the difference if any between cortisone injection versus bone marrow aspirate injection in the glenohumeral joint of patients with confirmed osteoarthritis. The investigators hope that results from a prospective randomized controlled pilot study on bone marrow aspirate (BMA) glenohumeral joint (GHJ) injections will provide valuable early information on an alternative treatment for GHJ osteoarthritis (OA). This novel study will also contribute clinical data to the growing pool of research around BMA in the treatment of osteoarthritis. This study has the potential to uncover a new and more effective therapy to add to the arsenal of an orthopaedic surgeon in the management of GHJ OA. This would provide improved care and treatment for those disabled by GHJ OA. Additionally, this knowledge would be applicable to a variety of medical practitioners who treat GHJ OA from the general orthopaedic surgeon to pain subspecialists.

DETAILED DESCRIPTION:
Glenohumeral joint (GHJ) osteoarthritis (OA) is a painful, progressive and debilitating condition that impairs quality of life. Currently, the only "cure" for arthritis is total joint replacement. This is a major operation that carries with it significant risks including infection, stiffness, limited range of motion, peri-prosthetic fracture and loosening. Furthermore, there are permanent post-operative restrictions, and in young or active people there is a significant rate of early revision surgery. Therefore, the goal of early shoulder OA management is symptom control, and postponement or prevention of the need for joint replacement.

Initial management options include physical therapy, pain-control medications, and intra-articular injections. Corticosteroid injections are the most commonly utilized injectables used in GHJ OA, with previous studies reporting good, short term pain relief and clinical improvement with corticosteroid injections for shoulder OA. However, corticosteroid injections may damage the collagen matrix of tendons and ligaments around the shoulder with repeated injections. Intra-articular hyaluronic acid (HA) injections have been proposed as an alternative to corticosteroid injections, and have demonstrated a clinically significant improvement in pain and function, albeit with a limited effect size.

Bone marrow aspirate concentrate (BMA) injections is a relatively recent option for the treatment of OA. BMA is a biological product that is produced through the centrifugation of the patient's own bone marrow, producing a cellular equivalent to iliac crest bone graft. This aspirate has been shown to contain, among other nucleated cells, mesenchymal stem cells (MSC's) and hematopoietic stem cells (which can directly convert to stromal MSC's).Furthermore, this minimally invasive procedure can be conducted as an outpatient procedure, saving operating room time.

Preliminary studies on intra-articular knee injections of BMA for early OA have reported statistically significant benefits in improved pain scores and function, with few adverse effects. The mechanism of action is likely through paracrine effects exerted by MSCs with the upshot being anti-inflammatory and potentially regenerative capabilities. These results are encouraging for the use of BMA in the shoulder, which is a non-weight bearing joint. Therefore, the investigators believe that the clinical improvements seen with BMA injections for knee OA will also be seen in the shoulder to an equal or greater extent.

To date there are no trials investigating injectable stem cell therapies in the shoulder. The investigators aim to conduct a randomized controlled study to test the safety and efficacy of BMA injections for the treatment of early to mid-stage GHJ OA.

1.2 Significance of Current Study

Results from a prospective randomized controlled pilot study on BMA GHJ injections will provide valuable early information on an alternative treatment for GHJ OA. This novel study will also contribute clinical data to the growing pool of research around BMA in the treatment of osteoarthritis.

This research group is proposing a randomized clinical trial prospectively comparing BMA GHJ injections versus Depo Medrol Cortisone GHJ injections. This study will include comprehensive clinical, functional and joint specific patient outcome scores.

After a comprehensive literature review, to the investigators knowledge, there are no studies on the efficacy of BMA injections for management of GHJ OA. Thus, this study will be the first to report on safety, efficacy and costs associated with BMA injections.

This innovative study has the potential to uncover a new and more effective therapy to add to the arsenal of an orthopaedic surgeon in the management of GHJ OA. This would provide improved care and treatment for people disabled by GHJ OA. Additionally, this knowledge would be applicable to a variety of medical practitioners who treat GHJ OA from the general orthopaedic surgeon to pain subspecialists.

ELIGIBILITY:
Inclusion Criteria:

* Men or women above the age of 18 - 65
* Primary diagnosis of glenohumeral joint osteoarthritis (Samilson and Prieto Stage 1, 2 or 3)
* Provision of informed consent

Exclusion Criteria:

* Prior condition (such as trauma, avascular necrosis, fracture, iatrogenic or chondrolysis) resulting in secondary osteoarthritis
* Previous surgical intervention for GHJ OA
* Previous injection of cortisone or other substance
* Inability to comply with rehabilitation or form completion
* Likely problems, in the judgement of the investigators, with maintaining follow-up (i.e. patients with no fixed address, patients not mentally competent to give consent, etc.)
* WSIB involvement
* Lawsuit involvement

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2015-10-08; Primary Completion 2020-07-30 (Actual); Study Completion 2021-11-23 (Actual)

PRIMARY OUTCOMES:
Western Ontario Osteoarthritis of the Shoulder (WOOS) Index | Survey administered at Baseline, and then change from baseline measured at 3 months post injection, 6 months post injection, and 12 months post injection with the survey being administered again at each of these time points.
  A 19 question, quality of life measurement tool for patients with osteoarthritis of the shoulder. WOOS assesses change in specific areas of daily life function from scores captured at pre injection baseline to those captured at 3, 6 and 12 month intervals.
  Patient responses are recorded with a mark placed on a scale by the patient for each of the 19 questions, with responses being measured quantitatively out of 100 per question, totaled per subsection (Physical Symptoms/600; Sports and Recreation/Work/500; Lifestyle/500;Emotions/300) , totaled out of 1900 overall. Marks placed at or near 0 on the scale indicate patient is not experiencing or affected by the symptom described in the question, while marks at or near 100 indicate the patient is very affected.
  Baseline survey completed on the day of the injection, repeated at 3, 6 and 12 months post injection to compare change in sub section score, and total score out of 1900 at the given time point, to the scores captured at baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Tim Dwyer, MBBS, PhD, Principal Investigator — Women's College Hospital
Locations (1):
- Women's College Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Levy JC, Virani NA, Frankle MA, Cuff D, Pupello DR, Hamelin JA. Young patients with shoulder chondrolysis following arthroscopic shoulder surgery treated with total shoulder arthroplasty. J Shoulder Elbow Surg. 2008 May-Jun;17(3):380-8. doi: 10.1016/j.jse.2007.11.004. Epub 2008 Mar 7. PMID 18329295
- [Background] Brander VA, Gomberawalla A, Chambers M, Bowen M, Nuber G. Efficacy and safety of hylan G-F 20 for symptomatic glenohumeral osteoarthritis: a prospective, pilot study. PM R. 2010 Apr;2(4):259-67. doi: 10.1016/j.pmrj.2010.02.010. PMID 20430327
- [Background] Millett PJ, Gobezie R, Boykin RE. Shoulder osteoarthritis: diagnosis and management. Am Fam Physician. 2008 Sep 1;78(5):605-11. PMID 18788237
- [Background] Silverstein E, Leger R, Shea KP. The use of intra-articular hylan G-F 20 in the treatment of symptomatic osteoarthritis of the shoulder: a preliminary study. Am J Sports Med. 2007 Jun;35(6):979-85. doi: 10.1177/0363546507300256. Epub 2007 Mar 29. PMID 17395958
- [Background] Merolla G, Sperling JW, Paladini P, Porcellini G. Efficacy of Hylan G-F 20 versus 6-methylprednisolone acetate in painful shoulder osteoarthritis: a retrospective controlled trial. Musculoskelet Surg. 2011 Dec;95(3):215-24. doi: 10.1007/s12306-011-0138-3. Epub 2011 May 13. PMID 21567154
- [Background] van der Windt DA, Koes BW, Deville W, Boeke AJ, de Jong BA, Bouter LM. Effectiveness of corticosteroid injections versus physiotherapy for treatment of painful stiff shoulder in primary care: randomised trial. BMJ. 1998 Nov 7;317(7168):1292-6. doi: 10.1136/bmj.317.7168.1292. PMID 9804720
- [Background] Colen S, Geervliet P, Haverkamp D, Van Den Bekerom MP. Intra-articular infiltration therapy for patients with glenohumeral osteoarthritis: A systematic review of the literature. Int J Shoulder Surg. 2014 Oct;8(4):114-21. doi: 10.4103/0973-6042.145252. PMID 25538430
- [Background] Wolfstadt JI, Cole BJ, Ogilvie-Harris DJ, Viswanathan S, Chahal J. Current concepts: the role of mesenchymal stem cells in the management of knee osteoarthritis. Sports Health. 2015 Jan;7(1):38-44. doi: 10.1177/1941738114529727. PMID 25553211
- [Background] Matsumoto T, Kawamoto A, Kuroda R, Ishikawa M, Mifune Y, Iwasaki H, Miwa M, Horii M, Hayashi S, Oyamada A, Nishimura H, Murasawa S, Doita M, Kurosaka M, Asahara T. Therapeutic potential of vasculogenesis and osteogenesis promoted by peripheral blood CD34-positive cells for functional bone healing. Am J Pathol. 2006 Oct;169(4):1440-57. doi: 10.2353/ajpath.2006.060064. PMID 17003498
- [Background] Matsumoto T, Mifune Y, Kawamoto A, Kuroda R, Shoji T, Iwasaki H, Suzuki T, Oyamada A, Horii M, Yokoyama A, Nishimura H, Lee SY, Miwa M, Doita M, Kurosaka M, Asahara T. Fracture induced mobilization and incorporation of bone marrow-derived endothelial progenitor cells for bone healing. J Cell Physiol. 2008 Apr;215(1):234-42. doi: 10.1002/jcp.21309. PMID 18205179
- [Background] Mifune Y, Matsumoto T, Kawamoto A, Kuroda R, Shoji T, Iwasaki H, Kwon SM, Miwa M, Kurosaka M, Asahara T. Local delivery of granulocyte colony stimulating factor-mobilized CD34-positive progenitor cells using bioscaffold for modality of unhealing bone fracture. Stem Cells. 2008 Jun;26(6):1395-405. doi: 10.1634/stemcells.2007-0820. Epub 2008 Apr 3. PMID 18388308
- [Background] Tondreau T, Meuleman N, Delforge A, Dejeneffe M, Leroy R, Massy M, Mortier C, Bron D, Lagneaux L. Mesenchymal stem cells derived from CD133-positive cells in mobilized peripheral blood and cord blood: proliferation, Oct4 expression, and plasticity. Stem Cells. 2005 Sep;23(8):1105-12. doi: 10.1634/stemcells.2004-0330. Epub 2005 Jun 13. PMID 15955825
- [Background] Centeno C, Pitts J, Al-Sayegh H, Freeman M. Efficacy of autologous bone marrow concentrate for knee osteoarthritis with and without adipose graft. Biomed Res Int. 2014;2014:370621. doi: 10.1155/2014/370621. Epub 2014 Sep 7. PMID 25276781
- [Background] Kim JD, Lee GW, Jung GH, Kim CK, Kim T, Park JH, Cha SS, You YB. Clinical outcome of autologous bone marrow aspirates concentrate (BMAC) injection in degenerative arthritis of the knee. Eur J Orthop Surg Traumatol. 2014 Dec;24(8):1505-11. doi: 10.1007/s00590-013-1393-9. Epub 2014 Jan 8. PMID 24398701
- [Background] Centeno CJ, Schultz JR, Cheever M, Robinson B, Freeman M, Marasco W. Safety and complications reporting on the re-implantation of culture-expanded mesenchymal stem cells using autologous platelet lysate technique. Curr Stem Cell Res Ther. 2010 Mar;5(1):81-93. doi: 10.2174/157488810790442796. PMID 19951252
- [Background] Peeters CM, Leijs MJ, Reijman M, van Osch GJ, Bos PK. Safety of intra-articular cell-therapy with culture-expanded stem cells in humans: a systematic literature review. Osteoarthritis Cartilage. 2013 Oct;21(10):1465-73. doi: 10.1016/j.joca.2013.06.025. Epub 2013 Jul 4. PMID 23831631
- [Background] Hendrich C, Franz E, Waertel G, Krebs R, Jager M. Safety of autologous bone marrow aspiration concentrate transplantation: initial experiences in 101 patients. Orthop Rev (Pavia). 2009 Oct 10;1(2):e32. doi: 10.4081/or.2009.e32. PMID 21808691
- [Background] Cole BJ, Schumacher HR Jr. Injectable corticosteroids in modern practice. J Am Acad Orthop Surg. 2005 Jan-Feb;13(1):37-46. doi: 10.5435/00124635-200501000-00006. PMID 15712981
- [Background] Kumar N, Newman RJ. Complications of intra- and peri-articular steroid injections. Br J Gen Pract. 1999 Jun;49(443):465-6. PMID 10562748
- [Background] Charalambous CP, Tryfonidis M, Sadiq S, Hirst P, Paul A. Septic arthritis following intra-articular steroid injection of the knee--a survey of current practice regarding antiseptic technique used during intra-articular steroid injection of the knee. Clin Rheumatol. 2003 Dec;22(6):386-90. doi: 10.1007/s10067-003-0757-7. Epub 2003 Oct 15. PMID 14677011
- [Background] Samilson RL, Prieto V. Dislocation arthropathy of the shoulder. J Bone Joint Surg Am. 1983 Apr;65(4):456-60. PMID 6833319